CLINICAL TRIAL: NCT06611020
Title: The Role of Adjuvant VaccInation After Conization for the Treatment for Cervical Dysplasia
Brief Title: Adjuvant VaccInation After Conization for the Treatment for CervicAL Dysplasia
Acronym: VITAL
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Valentina Chiappa, md, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: 570/20
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: HPV
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- treatment of HPV-related disease with or without vaccination

SUMMARY:
HPV vaccination has emerged as a strategy to reduce the risk of recurrence oafter excisional treatment. However, only few data are aviable. In this trial the investigators aim to assess the role of HPV vaccination in women traeted for HPV-related lesions

DETAILED DESCRIPTION:
Patients treated for HPV-related disease are counseled about the potential protective role of HPV vaccination. The investigators will monitor the risk of HPV recurrence in pateints who choce to have vaccination and who did not.

ELIGIBILITY:
Inclusion Criteria:

* Treatment of HPV-related disease

Exclusion Criteria:

* Previous HPV vaccination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pateints with HPV-related disease
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
HPV recurrence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Grazia Casadei, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided